CLINICAL TRIAL: NCT03092063
Title: Using Multifamily Groups to Improve Family-Centered Self-Management of Type 2 Diabetes Among Mexican-Americans
Brief Title: Using Multifamily Groups to Improve Self-Management of Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Alex Kopelowicz, M.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01NR015809 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-03-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Psychotherapy, Group

STUDY DESIGN:
Intervention Model Description: Diabetes Self-Management Education
Who Masked: Outcomes Assessor
Masking Description: Raters are blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tomando Control-Nurse (Experimental): Tomando Control de su Diabetes-Nurse is a culturally tailored, community-based, Diabetes Self-Management program delivered in a group format by licensed nurses working with individual patients and families.
  Interventions: Behavioral: Tomando Control-Nurse
- Tomando Control-Promotora (Experimental): Tomando Control de su Diabetes-Promotora is a culturally tailored, community-based, Diabetes Self-Management program delivered in a group format by community health workers (promotoras) working with individual patients and families.
  Interventions: Behavioral: Tomando Control-Promotora
- Enhanced Engagement-Nurse (Experimental): Tomando Control de su Diabetes-Nurse is a culturally tailored, community-based, Diabetes Self-Management program delivered in a group format by licensed nurses working with individual patients and families. If subjects do not benefit sufficiently, the subject may be randomized to receive three home visits to facilitate engagement with treatment.
  Interventions: Behavioral: Tomando Control-Nurse; Behavioral: Enhanced engagement
- Enhanced Engagement-Promotora (Experimental): Tomando Control de su Diabetes-Promotora is a culturally tailored, community-based, Diabetes Self-Management program delivered in a group format by licensed nurses working with individual patients and families. If subjects do not benefit sufficiently, the subject may be randomized to receive three home visits to facilitate engagement with treatment.
  Interventions: Behavioral: Tomando Control-Promotora; Behavioral: Enhanced engagement
- Multifamily Group-Promotora (Experimental): If subjects do not benefit sufficiently from the initial Tomando Control intervention offered by the promotoras, they may be randomized to receive a multifamily group intervention consisting of three components: three initial "joining" sessions conducted with each of the families separately; a one-day (six hour) educational workshop; and ongoing multifamily group sessions.
  Interventions: Behavioral: Tomando Control-Promotora; Behavioral: Multifamily Group
- Multifamily Group-Nurses (Experimental): If subjects do not benefit sufficiently from the initial Tomando Control intervention offered by the nurses, they may be randomized to receive a multifamily group intervention consisting of three components: three initial "joining" sessions conducted with each of the families separately; a one-day (six hour) educational workshop; and ongoing multifamily group sessions.
  Interventions: Behavioral: Tomando Control-Nurse; Behavioral: Multifamily Group

INTERVENTIONS:
Behavioral: Tomando Control-Nurse — Tomando Control de su Diabetes-Nurse is a community-based intervention given in six 2.5 hour sessions. The Spanish-language sessions are led by two trained Registered Nurses. Subjects covered in these sessions include: 1) techniques to deal with the symptoms of diabetes and associated conditions; 2) appropriate exercise; 3) healthy eating; 4) correct use of diabetes medications; and 5) working more effectively with health care providers in a collaborative partnership. Participants make weekly action plans, share experiences, and help each other solve problems they encounter in creating and carrying out their self-management strategies.
  Arms: Enhanced Engagement-Nurse; Multifamily Group-Nurses; Tomando Control-Nurse
Behavioral: Tomando Control-Promotora — Tomando Control de su Diabetes-Promotora is a community-based intervention given in six 2.5 hour sessions. The Spanish-language sessions are led by two trained promotoras. Subjects covered in these sessions include: 1) techniques to deal with the symptoms of diabetes and associated conditions; 2) appropriate exercise; 3) healthy eating; 4) correct use of diabetes medications; and 5) working more effectively with health care providers in a collaborative partnership. Participants make weekly action plans, share experiences, and help each other solve problems they encounter in creating and carrying out their self-management strategies.
  Arms: Enhanced Engagement-Promotora; Multifamily Group-Promotora; Tomando Control-Promotora
Behavioral: Enhanced engagement — The Tomando Control clinician (either a promotora or a Registered Nurse, depending on the original group assignment), will conduct up to three home visits that are designed to explain the purpose of the TC intervention to a key relative so as to re-engage the family member in the group process
  Arms: Enhanced Engagement-Nurse; Enhanced Engagement-Promotora
Behavioral: Multifamily Group — The multifamily group consists of three components: three initial "joining" sessions conducted with each of the families separately; a one-day (six hour) educational workshop; and ongoing multifamily group sessions.
  Arms: Multifamily Group-Nurses; Multifamily Group-Promotora

SUMMARY:
The overall objective of this study is to construct an adaptive intervention that integrates family members and patients as partners in care while promoting diabetes self-management for Mexican Americans with Type 2 diabetes. The project incorporates four evidence-based, culturally tailored treatments using a Sequential, Multiple Assignment Randomized Trial to help determine what sequence of intervention strategies work most efficiently and for whom.

DETAILED DESCRIPTION:
The project evaluates four culturally adapted, family-based treatments designed to improve health status, self-management behaviors and self-efficacy among Mexican-Americans with Type 2 diabetes using a Sequential, Multiple Assignment Randomized Trial in a public health setting. In the first phase of the study, subjects will be randomly assigned to six 2.5 hour sessions (three months) of either: 1) Tomando Control de su Diabetes (TC), a culturally tailored, community-based, Diabetes Self-Management program delivered in a group format by community health workers (promotoras) working with individual patients and families; or 2) TC delivered by health professionals (licensed nurses). Evaluations will be made at baseline, three months, six months and 12 months. After six weeks of treatment (at the midway point of the intervention), subjects will be assessed for improvement in diabetes self-management behaviors (the primary outcome). In the second phase of the study, those subjects who have improved their diabetes self-management behaviors by 50% over baseline will be continued in their assigned treatment for the duration of three months. Those subjects who do not meet this target will be re-randomized to receive either: 1) an augmented version of TC that has a specific focus on engaging family members; or 2) a multifamily group treatment led by nurses specially trained in teaching diabetes self-management skills for an additional three months.

ELIGIBILITY:
Inclusion Criteria:

1. Mexican origin and speaks Spanish fluently
2. age 18 years or older
3. medical chart diagnosis of Type 2 diabetes
4. living with at least one adult family member who is willing to participate.

Exclusion Criteria:

1. diagnosis of Type 1 diabetes
2. participation in another Diabetes Self-management education program within the past 12 months
3. pregnancy
4. significant cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Self-Management Behaviors (Revised Summary of Diabetes Self-Care Activities) | This outcome measure will be assessed at baseline, six weeks, three months, six months and 12 months. The primary outcome is change from baseline as compared to the subsequent assessment points.
  This 11-item scale assesses ADA-recommended health activities in diet, exercise, glucose self-monitoring, medication adherence and foot care. The mean number of days in the past week that activities are performed is calculated on a scale of 0-7; a high mean score indicates better diabetes self-management.

SECONDARY OUTCOMES:
Diabetes Self-Efficacy (Stanford Self-Efficacy Scale) | This outcome measure will be assessed at baseline, three months, six months and 12 months.
  An 8-item measure that assesses the confidence of a person with diabetes to manage diet, exercise, knowledge of blood glucose and the illness, and control over diabetes. Scores range from 1-10, from no confidence to totally confident; higher scores indicate greater confidence.
Diabetes knowledge (Spoken Knowledge in Low Literacy Patients with Diabetes scale) | This outcome measure will be assessed at baseline, three months, six months and 12 months.
  This 10-item scale assesses knowledge of glucose management, lifestyle modifications, recognition and treatment of hyper- and hypoglycemia, and activities to prevent long-term consequences of the disease. Correct answers receive a score of 1. Each item score is summed ranging from 0-10, with a high score indicating better knowledge about diabetes.
Family Support (Diabetes Family Support Behavior Checklist) | This outcome measure will be assessed at baseline, three months, six months and 12 months.
  This 17-item scale uses a 5-point Likert range to assess perceptions of family member support of the person with T2DM in medication taking, glucose self-monitoring, exercise and diet. Positive and negative items are summed separately and higher scores indicate stronger perception of family support.
Collaborative goal setting (Patient Assessment of Chronic Illness Care) | This outcome measure will be assessed at baseline, three months, six months and 12 months.
  A 20-item patient survey that evaluates the quality and patient centeredness of chronic illness care received according to the Chronic Care Model paradigm. The questionnaire is divided into five subscales to reflect the key components of the Chronic Care Model: patient activation, delivery system design & decision support, goal setting & tailoring, problem-solving & contextual, and follow-up/coordination. Each item has a score from 1 (never) to 5 (always). Patients self-report how often they received specific types of medical care during the past six months.
Glycemic control | This outcome measure will be assessed at baseline, three months, six months and 12 months.
  Hemoglobin A1c serum level

CONTACTS AND LOCATIONS:
Overall Officials: alex kopelowicz, MD, Principal Investigator — Olive View-UCLA Education & Research Institute
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kopelowicz A, Wali S, Polzin R, Ruiz ME, Nandy K. Promotore-Led Versus Registered Nurse-Led Diabetes Self-Management Education in Mexican Americans: A Randomized Clinical Trial. Sci Diabetes Self Manag Care. 2023 Oct;49(5):374-383. doi: 10.1177/26350106231192353. Epub 2023 Aug 18. PMID 37593833
- [Derived] Kopelowicz A, Nandy K, Ruiz ME, Polzin R, Kurator K, Wali S. Improving Self-management of Type 2 Diabetes in Latinx Patients: Protocol for a Sequential Multiple Assignment Randomized Trial Involving Community Health Workers, Registered Nurses, and Family Members. JMIR Res Protoc. 2023 Jan 16;12:e44793. doi: 10.2196/44793. PMID 36645708